CLINICAL TRIAL: NCT03376074
Title: Interest of Oxygenated Hypothermic Perfusion in Preservation of Hepatic Grafts From Expanded Criteria Donors. A Prospective Monocentric Study.
Brief Title: Interest of Oxygenated Hypothermic Perfusion (PHO) in Preservation of Hepatic Grafts From Expanded Criteria Donors
Acronym: PERPHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC16_9792_PERPHO; 2017-A00085-48 (Other: ID-RCB number)
Record Dates: First submitted 2017-12-07; First posted 2017-12-18 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Injury
Keywords: liver transplantation; hypothermic machine liver perfusion; extended criteria liver grafts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypothermic oxygenated perfusion (HOPE) (Experimental): Application of HOPE for 2 hours
  Interventions: Device: Hypothermic oxygenated perfusion (HOPE)
- Conventional cold storage (Active Comparator)
  Interventions: Other: Conventional cold storage

INTERVENTIONS:
Device: Hypothermic oxygenated perfusion (HOPE) — 25 patients: Application of HOPE for 2 hours, perfusion rate 100-150 ml/min, pressure controlled, perfusion pressure < 3 mm Hg, perfusion route portal vein, recirculating system, perfusion volume 2 L, perfusate solution (UWMP®), perfusate temperature 4-12 °C, perfusate oxygenation 40 KPa
  Arms: Hypothermic oxygenated perfusion (HOPE)
Other: Conventional cold storage — 75 patients transplanted in Rennes between 2010 and 2015 with a cold stored grafts, matched (ratio 1: 3) using a propensity score calculated according to some parameters
  Arms: Conventional cold storage

SUMMARY:
Interest of oxygenated hypothermic perfusion in preservation of hepatic grafts from expanded criteria donors.

DETAILED DESCRIPTION:
The excellent results of liver transplantation (LT) have led to a significant increase in the number of patients awaiting transplantation. At the same time, the number of grafts remains stable. To extend the donor pool, the use of Extended Criteria Donor (ECD) donors graft increased each year despite the fact that these graft are known to be more vulnerable to ischemia-reperfusion injuries induced by cold storage preservation (CS). Their use is therefore associated with a greater risk of postoperative dysfunction of the graft. This risk can be reduced by improving preservation quality.

The preservation by hypothermic oxygenated perfusion (HOPE) consists of keeping the graft in hypothermia (4 to 12 °C) on an machine perfusion (MP) using a specific solution, saturated with oxygen. In kidney transplantation, the use of MP has been shown to improve graft function as well as graft survival, especially for ECD grafts.

In liver transplantation, experimental studies on animal models have demonstrated the superiority of HOPE over CS regarding graft function and survival. These results have been confirmed in humans on small retrospective series.

As HOPE is an expensive procedure, obtaining evidence of its effectiveness could result in a reimbursement of the additional cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Candidates for a first orthotopic liver transplantation, without transplantation of another associated organ (kidney, pancreas, heart, lung, intestine)
* With cirrhosis whatever its etiology and gravity
* With or without hepatocarcinoma
* Having given free, informed and written consent
* LT made from a whole graft, harvested from a brain-dead donor with ECD criteria, defined as the presence of at least one of the following criteria:

  * Age> 65 years
  * BMI> 30 kg / m2
  * Duration of hospitalization in intensive care unit> 7 days
  * Natremia> 155 mmol / l
  * AST> 150 IU / ml
  * ALT> 170 IU / ml
  * Occurrence of cardiac arrest before harvesting
  * Macrovacuolar steatosis> 30% on liver histology

Exclusion Criteria:

* History of organ transplantation
* Transplantation in emergency
* Transplantation from a living donor, a reduced graft or a graft from a deceased donor by cardiac arrest (DCD)
* Major persons subject to legal protection (safeguard of justice, guardianship), persons deprived of their liberty

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the performance of HOPE in the preservation of ECD liver grafts on graft function recovery | Day 7
  Occurrence of early allograft dysfunction and / or primary non function

SECONDARY OUTCOMES:
Evaluation of the impact of PHO during the conservation of ECD liver grafts on intraoperative morbidity | Day 1
  Number of intraoperative transfusions
Evaluation of the impact of PHO during the conservation of ECD liver grafts on intraoperative morbidity | Day 1
  Incidence of reperfusion syndrome defined as a 30 % decrease of mean arterial pressure, for at least 1 minute, during the 5 minutes following revascularization
Evaluation of the impact of PHO during the conservation of ECD liver grafts on postoperative morbidity | Day 7
Evaluation of graft's survival | Month 3
  Occurrence of a vascular and biliary complication
Number of days of hospitalization (initial stay) after transplantation | Postoperative course
Number of days of hospitalization after transplantation | Month 3
Cost of the initial stay | Postoperative course
Cost of the hospitalization stay | Month 3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rayar M, Beaurepaire JM, Bajeux E, Hamonic S, Renard T, Locher C, Desfourneaux V, Merdrignac A, Bergeat D, Lakehal M, Sulpice L, Houssel-Debry P, Jezequel C, Camus C, Bardou-Jacquet E, Meunier B. Hypothermic Oxygenated Perfusion Improves Extended Criteria Donor Liver Graft Function and Reduces Duration of Hospitalization Without Extra Cost: The PERPHO Study. Liver Transpl. 2021 Feb;27(3):349-362. doi: 10.1002/lt.25955. PMID 33237618